CLINICAL TRIAL: NCT06320470
Title: MIVetsCan: Cannabis Coaching for Veteran Pain Management Trial (Phase 1)
Brief Title: MIVetsCan: Can-Coach Trial (Phase 1)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Michigan, State of, Licensing and Regulatory Affairs (Unknown)
Responsible Party: Principal Investigator, Kevin Boehnke, Research Assistant Professor, Anesthesiology, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HUM00231159a; VMR2022-03 (Other Grant/Funding Number: Michigan, State of, Licensing and Regulatory Affairs, Department of 573000)
Record Dates: First submitted 2024-02-21; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Chronic Pain
Keywords: Veteran; Cannabis
MeSH Terms: conditions — Chronic Pain; Marijuana Abuse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Education (Experimental): Prior to the educational sessions, study participants will be given access to educational materials (e.g., handouts, videos) that provide an overview of information regarding cannabis products, effects, and pain. These materials will be developed with insight from the study team and the Community Advisory Board.
  Educational content will include known side effects of cannabis (e.g., common effects like dizziness or sedation, rare side effects like hallucinations or vomiting) as well as specific risks associated with administration routes, such as respiratory harm from smoking or unregulated vaporized concentrate products, and the delayed onset of edible products. Sessions will help the participants appropriately select products for use.
  Interventions: Behavioral: Educational Session

INTERVENTIONS:
Behavioral: Educational Session — The initial session will last about 45 to 60 minutes. The subsequent 3 sessions are anticipated to take about 20-30 minutes.

SUMMARY:
The goal of the MIVetsCan Can-Coach Trial is to pilot and modify a trial of four coaching sessions to help Veterans with chronic pain use their own cannabis products more effectively to manage pain and related symptoms.

DETAILED DESCRIPTION:
All study interactions will be done virtually and recruitment data is exploratory.

ELIGIBILITY:
Inclusion Criteria:

* United States Veteran
* Experiencing chronic pain (pain lasting 3 or more months)
* Worst pain of ≥3 out of 10 using a 0-10 Numeric Rating Scale (NRS)
* Are planning or currently using cannabidiol (CBD) or cannabis products for pain management
* Able to read and speak English sufficiently to allow for informed consent and active participation in the educational intervention sessions
* Willingness to attend all study visits (conducted virtually)
* Willingness to fill out periodic assessments via smartphone to assess symptom status and cannabis use (protocol has more details)

Exclusion Criteria:

* Inability to provide informed consent (e.g., cognitive impairment, unable to sufficiently communicate in English)
* Participant states participant is pregnant
* Current diagnosis or past history of a psychotic disorder (schizophrenia spectrum, except substance/medication -induced or due to another condition)
* Current diagnosis or past history of bipolar disorder
* Unable to attend study visits
* Risk for eminent harm - Suicidal ideation or wish to die as assessed with the Positive and Negative Suicide Ideation (PANSI) questionnaire and further risk assessment by study team members
* Any impairment, activity, behavior, or situation that in the judgment of the study team would prevent satisfactory completion of the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Patient Global Impression of Change (PGIC) score | Week 14
  Patient's Global Impression of Change (PGIC) scale will be used. This is a 7 point scale ranging from 1 (very much worse) to 7 (very much better).

SECONDARY OUTCOMES:
Average satisfaction level of the cannabis coaching overall assessed from a single survey question on satisfaction. | Following intervention, up to approximately Week 14
  Self-report during the end of treatment survey, from not at all satisfied (1), somewhat satisfied (2), satisfied (3), very satisfied (4), completely satisfied (5).
Average helpfulness level of the cannabis coaching assessed from a single survey question on cannabis coaching. | Following intervention, up to approximately Week 14
  Measured from self-report during the end of treatment survey, from not at all helpful (1), somewhat helpful (2), helpful (3), very helpful (4), completely helpful (5).

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Boehnke, PhD, Study Chair — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boehnke KF, Bowyer G, McAfee J, Smith T, Klida C, Kurtz V, Litinas E, Purohit P, Arewasikporn A, Horowitz D, Thomas L, Eckersley J, Railing M, Williams DA, Clauw DJ, Kidwell KM, Bohnert ASB, Bergmans RS. Feasibility pilot of a novel coaching intervention to optimize cannabis use for chronic pain management among Veterans. J Cannabis Res. 2025 Jan 25;7(1):7. doi: 10.1186/s42238-025-00265-z. PMID 39856785